CLINICAL TRIAL: NCT04191499
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Inavolisib Plus Palbociclib and Fulvestrant Versus Placebo Plus Palbociclib and Fulvestrant in Patients With PIK3CA-Mutant, Hormone Receptor-Positive, HER2-Negative, Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Inavolisib + Palbociclib + Fulvestrant vs Placebo + Palbociclib + Fulvestrant in Participants With PIK3CA-Mutant, Hormone Receptor-Positive, HER2-Negative, Locally Advanced or Metastatic Breast Cancer
Acronym: INAVO120
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO41554; 2019-002455-42 (EudraCT Number); 2023-505812-39-00 (EU CTIS Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; palbociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inavolisib + Palbociclib + Fulvestrant (Experimental): Participants will receive inavolisib, palbociclib, and fulvestrant.
  Interventions: Drug: Inavolisib; Drug: Palbociclib; Drug: Fulvestrant
- Placebo + Palbociclib + Fulvestrant (Placebo Comparator): Participants will receive placebo, palbociclib, and fulvestrant. Participants randomized to the placebo arm who are still deriving benefit from the study treatment will be given an optional opportunity to crossover to the inavolisib arm.
  Interventions: Drug: Placebo; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Inavolisib — Participants will receive oral inavolisib on Days 1-28 of each 28-day cycle.
  Other Names: GDC-0077
  Arms: Inavolisib + Palbociclib + Fulvestrant
Drug: Placebo — Participants will receive oral placebo on Days 1-28 of each 28-day cycle.
  Arms: Placebo + Palbociclib + Fulvestrant
Drug: Palbociclib — Participants will receive oral palbociclib on Days 1-21 of each 28-day cycle.
Drug: Fulvestrant — Participants will receive intramuscular (IM) fulvestrant approximately every 4 weeks.

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of inavolisib in combination with palbociclib and fulvestrant compared with placebo plus palbociclib and fulvestrant in participants with PIK3CA-mutant, hormone receptor (HR)-positive, HER2-negative locally advanced or metastatic breast cancer whose disease progressed during treatment or within 12 months of completing adjuvant endocrine therapy and who have not received prior systemic therapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of HR+/HER2- breast cancer
* Metastatic or locally advanced disease not amenable to curative therapy
* Progression of disease during adjuvant endocrine treatment or within 12 months of completing adjuvant endocrine therapy with an aromatase inhibitor or tamoxifen
* Receiving LHRH agonist therapy for at least 2 weeks prior to Day 1 of Cycle 1 if pre/peri-menopausal
* Confirmation of biomarker eligibility (detection of specified mutation(s) of PIK3CA via specified test)
* Consent to provide fresh or archival tumor tissue specimen
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1); evaluable "bone-only" disease is not eligible; "bone-only" disease with at least one measurable, soft-tissue component, even if considered disease that is limited to bone but has lytic or mixed lytic/blastic lesions and at least one measurable soft-tissue component per RECIST v1.1 may be eligible
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Life expectancy of > 6 months
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment

Exclusion Criteria

* Metaplastic breast cancer
* Any history of leptomeningeal disease or carcinomatous meningitis
* Any prior systemic therapy for metastatic breast cancer
* Prior treatment with fulvestrant or any selective estrogen-receptor degrader, with the exception of participants that have received fulvestrant or any selective estrogen-receptor degrader as part of neoadjuvant therapy only and with treatment duration of no longer than 6 months
* Prior treatment with any PI3K, AKT, or mTOR inhibitor, or any agent whose mechanism of action is to inhibit the PI3K-AKT-mTOR pathway
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Known and untreated, or active CNS metastases. Patients with a history of treated CNS metastases may be eligible
* Active inflammatory or infectious conditions in either eye, or any eye conditions expected to require surgery during the study treatment period
* Symptomatic active lung disease, or requiring daily supplemental oxygen
* History of inflammatory bowel disease or active bowel inflammation
* Anti-cancer therapy within 2 weeks before study entry
* Investigational drug(s) within 4 weeks before randomization
* Prior radiotherapy to >= 25% of bone marrow, or hematopoietic stem cell or bone marrow transplantation
* Chronic corticosteroid therapy or immunosuppressants
* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or within 2 weeks after the final dose of study treatment
* Major surgical procedure, or significant traumatic injury, within 28 days prior to Day 1 of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2027-11-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (135):
- United States (10):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Massachusetts General Hospital., Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (3):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
  - Hosp Provincial D. Centenarios, Rosario
- Australia (6):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Western Health, Fitzroy, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - London Regional Cancer Program, London Health Sciences Centre, Baines Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital du Saint Sacrement, Québec, Quebec
- China (13):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Fudan University Shanghai Cancer Center, Shanghai
  - Hebei Medical University Fourth Hospital, Shijiazhuang
  - Tianjin Cancer Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Vejle Sygehus, Vejle, Denmark
- France (6):
  - Centre Jean Perrin Centre Regional de Lutte Contre Le Cancer D auvergne, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hopital Prive Jean Mermoz, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
- Georgia (2):
  - Israel-Georgian Medical Research Clinic Healthycore, Tbilisi
  - Tbilisi Oncology Dispensary, Tbilisi
- Germany (6):
  - Ambulantes Tumorzentrum Spandau, Berlin
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH, Trier
  - Universitätsfrauenklinik Ulm, Ulm
- Greece (4):
  - Anticancer Hospital Ag. Savas, Athens
  - Univ General Hosp Heraklion, Heraklion
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Italy (5):
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - Az. Osp. Spedali Civili, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Malaysia (3):
  - National Cancer Institute IKN, Putrajaya, Federal Territory of Putrajaya
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Sarawak General Hospital, Sarawak, Sarawak
- Palmerston North Hospital, Palmerston North, New Zealand
- Poland (3):
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
- Portugal (2):
  - Centro Clinico Champalimaud, Lisbon
  - IPO do Porto, Porto
- Russia (7):
  - Moscow Clinical Scientific Center, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center, Moscow, Moscow Oblast
  - LLC Medscan, Moskva, Moscow Oblast
  - Clinical Hospital Lapino (LLC Haven), Yudino, Moscow Oblast
  - Medical Clinic "AB Medical group", Saint Petersburg, Sankt-Peterburg
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncology Hospital, Yaroslavl
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (11):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital del Mar, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Insituto Catalán de Oncologia (ICO), Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (5):
  - Kaohsiung Medical Uni Chung-Ho Hospital, Kaohsiung City
  - Veterans General Hospital, Taipei
  - National Taiwan Uni Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Tri-Service General Hospital, Division of General Surgery, Taipei
- Thailand (4):
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Chulabhorn Hospital, Lak Si
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (5):
  - Adana Baskent University Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Ege University Medical Faculty, Bornova, ?zm?r
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital, Istanbul
- Ukraine (6):
  - SI Institute of general&urgent surgery n/a Zaytseva V.T NAMSU, Kharkiv, Kharkiv Governorate
  - Municipal Institution SubCarpathian Clinical Oncological Centre, Ivano-Frankivsk, KIEV Governorate
  - Uzhhorod Central City Clinical Hospital, Uzhhorod, KIEV Governorate
  - City Clinical Hospital #4, Dnipropetrovsk
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council, Kryvyi Rih
  - Kyiv City Clinical Oncological Center, Kyiv
- United Kingdom (4):
  - Royal Marsden Hospital - Fulham, London
  - Mount Vernon Hospital, Northwood
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Jhaveri KL, Im SA, Saura C, Loibl S, Kalinsky K, Schmid P, Loi S, Thanopoulou E, Shankar N, Jin Y, Stout TJ, Clark TD, Song C, Juric D, Turner NC. Overall Survival with Inavolisib in PIK3CA-Mutated Advanced Breast Cancer. N Engl J Med. 2025 Jul 10;393(2):151-161. doi: 10.1056/NEJMoa2501796. Epub 2025 May 31. PMID 40454641
- [Derived] Turner NC, Im SA, Saura C, Juric D, Loibl S, Kalinsky K, Schmid P, Loi S, Sunpaweravong P, Musolino A, Li H, Zhang Q, Nowecki Z, Leung R, Thanopoulou E, Shankar N, Lei G, Stout TJ, Hutchinson KE, Schutzman JL, Song C, Jhaveri KL. Inavolisib-Based Therapy in PIK3CA-Mutated Advanced Breast Cancer. N Engl J Med. 2024 Oct 31;391(17):1584-1596. doi: 10.1056/NEJMoa2404625. PMID 39476340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 123 investigative centers in 28 countries. This study is still ongoing.
Pre-assignment Details: A total of 325 participants with phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit, alpha isoform (PIK3CA) mutation, hormone receptor-positive, human epidermal growth factor receptor 2 negative (HER2-) locally advanced or metastatic breast cancer were randomized in 1:1 ratio to Inavolisib+ Palbociclib + Fulvestrant (Inavo+Palbo+Fulv) arm or Placebo + Palbociclib + Fulvestrant (Pbo+Palbo+Fulv) arm in this study.
Groups:
- Inavo+Palbo+Fulv: Participants received inavolisib, 9 milligrams (mg), orally, once daily (QD) on Days 1-28 of each 28 day cycle along with palbociclib 125 mg, orally, QD on Days 1-21 and fulvestrant, 500 mg, intramuscular (IM) injections on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent 28 day cycle until unequivocal disease progression, unacceptable toxicity, participant withdrawal of consent, or study termination.
- Pbo+Palbo+Fulv: Participants received placebo, orally, QD on Days 1-28 of each 28 day cycle along with palbociclib 125 mg, orally, QD on Days 1-21 and fulvestrant, 500 mg, IM injections on Days 1 and 15 of Cycle 1 and then of Day 1 of each subsequent 28 day cycle until unequivocal disease progression, unacceptable toxicity, participant withdrawal of consent, or study termination.
Period: Overall Study
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv
Started | 161 | 164
Completed | 0 | 0
Not Completed | 161 | 164
Not completed — Adverse Event | 1 | 0
Not completed — Death | 42 | 55
Not completed — Lost to Follow-up | 4 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive Disease | 1 | 0
Not completed — Symptomatic Deterioration | 1 | 0
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Ongoing in the study | 104 | 97

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to receive the treatment they were assigned.
Groups:
- Inavo+Palbo+Fulv: Participants received inavolisib, 9 mg, orally, QD on Days 1-28 of each 28 day cycle along with palbociclib 125 mg, orally, QD on Days 1-21 and fulvestrant, 500 mg, IM injections on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent 28 day cycle until unequivocal disease progression, unacceptable toxicity, participant withdrawal of consent, or study termination.
- Total: Total of all reporting groups
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv | Total
Number analyzed (Participants) | 161 | 164 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.9) | 54.1 (11.2) | 54.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 163 | 319
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 145 | 149 | 294
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 61 | 63 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 94 | 97 | 191
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 or death from any cause (whichever occurs first). Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions was also considered progression. Data for participants without the occurrence of PD or death as of the clinical cutoff date (CCOD) were censored at the time of the last tumor assessment prior to the CCOD. Median PFS was calculated using the Kaplan-Meier methodology.
Time Frame: Up to 3.7 years
Population: FAS included all participants who were randomized to receive the treatment they were assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv
Number analyzed (Participants) | 161 | 164
months | 15 [11.3 to 20.5] | 7.3 [5.6 to 9.3]
Statistical Analysis 1: Comparison: Inavo+Palbo+Fulv vs Pbo+Palbo+Fulv; Hazard ratios were estimated by Cox regression. Hazard ratios and log-rank p-values are using stratified methods by stratifying Visceral Disease, Endocrine Resistance, and Region; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.32 to 0.59]

2. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a complete response (CR) and/or partial response (PR) on at least two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR is defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum in the study (nadir), including baseline.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

3. Secondary Outcome: Percentage of Participants With Best Overall Response Rate (BOR)
Description: BOR is defined as the percentage of participants with a CR or PR, as determined by the investigator according to RECIST v1.1. CR is defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum in the study (nadir), including baseline.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first occurrence of a CR or PR to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1, or death from any cause (whichever occurs first). CR is defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum in the study (nadir), including baseline. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

5. Secondary Outcome: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with a CR, PR, and/or stable disease (SD) for at least 24 weeks, as determined by the investigator according to RECIST v1.1. CR= disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the smallest sum in the study (nadir), including baseline. PD=at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum in the study.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

7. Secondary Outcome: Time to Deterioration (TTD) in Pain
Description: TTD in pain is defined as the time from randomization to the first documentation of a ≥ 2-point increase from baseline on the "worst pain" item from the Brief Pain Inventory-Short Form (BPI-SF). BPI-SF is a self-administered questionnaire in which the participant was asked to rate severity on a 10-point scale where 0 represents 'No pain/No interference' and 10 represents 'Pain/Interference as bad as you can imagine'. A ≥2-point change is defined as clinically meaningful difference.
Time Frame: From randomization to first documentation of a ≥ 2-point increase (Up to approximately 6 years)
Reporting Status: Not Posted, anticipated posting 2031-09

8. Secondary Outcome: TTD in Physical Function (PF)
Description: TTD in physical function is defined as the time from randomization to the first documentation of a ≥ 10-point decrease from baseline held for two consecutive cycles or initial decrease followed by death or treatment discontinuation within three weeks of last assessment in the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) PF scale (items 1-5). A ≥10-point change is defined as a clinically meaningful difference. EORTC QLQ-C30 is a cancer-specific health-related quality-of life (QoL) questionnaire with 30 questions. For the PF scale, participant responses to 5 questions about daily activities (strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves, or using the toilet) is scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score indicating worst functioning.
Time Frame: Treatment: Day 1 of Cycles 1-3, then Day 1 of every other cycle until treatment discontinuation. Post-treatment: Every 8 weeks for 2 years, then every 12 weeks thereafter, to end of study (up to 6 years) (Cycle length = 28 days)]
Reporting Status: Not Posted, anticipated posting 2031-09

9. Secondary Outcome: TTD in Role Function (RF)
Description: TTD in Role Function is defined as the time from randomization to the first documentation of a ≥ 10-point decrease from baseline held for two consecutive cycles, or initial decrease followed by death or treatment discontinuation within three weeks of last assessment in the EORTC QLQ-C30 RF scale (items 6 and 7). A ≥10-point change is defined as clinically meaningful difference. EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. For the role functioning scale, participant responses to the 2 questions "Q6: Were you limited in doing either your work or daily activities" and "Q7: Were you limited in pursuing your hobbies or other leisure time activities" were scored on a 4-point scale (1=Not at All to 4=Very Much). The scores were linearly transformed on a scale of 0 to 100, with a low score indicating better functioning.
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2031-09

10. Secondary Outcome: TTD in Global Health Status (GHS)
Description: TTD in (GHS)/health-related quality of life (HRQoL) is defined as the time from randomization to the first documentation of a ≥ 10-point decrease from baseline held for two consecutive cycles, or initial decrease followed by death or treatment discontinuation within three weeks of last assessment in the EORTC QLQ-30 GHS/HRQoL scale. A ≥10-point change is defined as clinically meaningful difference. EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. Participant responses to the questions regarding Global Health Status (Q29: GHS; "How would you rate your overall health during the past week?") and Quality of Life (Q30: QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better outcome.
Time Frame: as for outcome 8
Reporting Status: Not Posted, anticipated posting 2031-09

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is an untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product.
Time Frame: Up to approximately 6 years
Reporting Status: Not Posted, anticipated posting 2031-09

12. Secondary Outcome: Plasma Concentration of Inavolisib
Time Frame: Predose on Cycle 1 Days 1, 8 and 15 and Cycle 2 Day 15; 3 hours post-dose on Cycle 1 Days 1 and 15 (Cycle length = 28 days)
Population: Pharmacokinetic (PK) evaluable population included all participants who received at least one dose of study drug, had at least one post-baseline sample, and was based on the treatment participants actually received. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Inavo+Palbo+Fulv
Number analyzed (Participants) | 151
nanogram/milliliter (ng/ml)
  Predose, Cycle 1 Day 1 | NA (NA) — The data was not estimable as the samples were below the lower limit of quantification (BLLQ).
  3 hours Post-dose, Cycle 1 Day 1 | 36 (223)
  Predose, Cycle 1 Day 8: number analyzed (Participants) | 121
  Predose, Cycle 1 Day 8 | 17.8 (134)
  Predose, Cycle 1 Day 15: number analyzed (Participants) | 117
  Predose, Cycle 1 Day 15 | 13.6 (240)
  3 hours Post-dose, Cycle 1 Day 15: number analyzed (Participants) | 120
  3 hours Post-dose, Cycle 1 Day 15 | 59.2 (119)
  Predose, Cycle 2 Day 15: number analyzed (Participants) | 115
  Predose, Cycle 2 Day 15 | 16.9 (124)

13. Secondary Outcome: Plasma Concentration of Palbociclib
Time Frame: as for outcome 12
Population: PK evaluable population included all participants who received at least one dose of study drug, had at least one post-baseline sample, and was based on the treatment participants actually received. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv
Number analyzed (Participants) | 154 | 153
ng/ml
  Predose, Cycle 1 Day 1 | NA (NA) — The data was not estimable as the samples were BLLQ. | NA (NA) — The data was not estimable as the samples were BLLQ.
  3 hours Post-dose, Cycle 1 Day 1 | 20.7 (182) | 22.9 (251)
  Predose, Cycle 1 Day 8: number analyzed (Participants) | 134 | 138
  Predose, Cycle 1 Day 8 | 73.9 (56) | 74.5 (50)
  Predose, Cycle 1 Day 15: number analyzed (Participants) | 136 | 134
  Predose, Cycle 1 Day 15 | 69.9 (78) | 73.3 (65)
  3 hours Post-dose, Cycle 1 Day 15: number analyzed (Participants) | 138 | 131
  3 hours Post-dose, Cycle 1 Day 15 | 96.7 (55) | 98.0 (62)
  Predose, Cycle 2 Day 15: number analyzed (Participants) | 130 | 122
  Predose, Cycle 2 Day 15 | 58.5 (111) | 66.9 (90)

14. Secondary Outcome: Plasma Concentration of Fulvestrant
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv
Number analyzed (Participants) | 154 | 154
ng/ml
  Predose, Cycle 1 Day 1 | NA (NA) — The data was not estimable as the samples were BLLQ. | NA (NA) — The data was not estimable as the samples were BLLQ.
  3 hours Post-dose, Cycle 1 Day 1 | 1.03 (200) | 0.815 (200)
  Predose, Cycle 1 Day 8: number analyzed (Participants) | 137 | 137
  Predose, Cycle 1 Day 8 | 17.5 (46) | 16.2 (46)
  Predose, Cycle 1 Day 15: number analyzed (Participants) | 138 | 142
  Predose, Cycle 1 Day 15 | 11.9 (37) | 10.9 (42)
  3 hours Post-dose, Cycle 1 Day 15: number analyzed (Participants) | 139 | 139
  3 hours Post-dose, Cycle 1 Day 15 | 12.2 (44) | 11.1 (43)
  Predose, Cycle 2 Day 15: number analyzed (Participants) | 137 | 132
  Predose, Cycle 2 Day 15 | 18.0 (37) | 17.3 (37)

ADVERSE EVENTS:
Time Frame: Up to 3.7 years
Description: Safety analysis set (SAS) included all participants who were exposed to study treatment. 2 participants randomized to the Pbo+Palbo+Fulv arm received at least one dose of inavolisib in error and were included in the Inavo+Palbo+Fulv arm in SAS population for the purposes of safety analyses. This study is ongoing, and data collected up to the primary completion date are reported here.
Arm/Group | Inavo+Palbo+Fulv | Pbo+Palbo+Fulv
All-Cause Mortality (participants affected / at risk) | 43/162 | 54/162
Serious Adverse Events (participants affected / at risk) | 39/162 | 17/162
Other Adverse Events (participants affected / at risk) | 157/162 | 158/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inavo+Palbo+Fulv (N=162) | Pbo+Palbo+Fulv (N=162)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inavo+Palbo+Fulv (N=162) | Pbo+Palbo+Fulv (N=162)
Anaemia (Blood and lymphatic system disorders) | 58 (102) | 59 (104)
Leukopenia (Blood and lymphatic system disorders) | 28 (81) | 40 (80)
Neutropenia (Blood and lymphatic system disorders) | 88 (251) | 89 (215)
Thrombocytopenia (Blood and lymphatic system disorders) | 36 (95) | 41 (65)
Dry eye (Eye disorders) | 14 (14) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 16 (20) | 10 (15)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16) | 11 (13)
Constipation (Gastrointestinal disorders) | 24 (35) | 23 (27)
Diarrhoea (Gastrointestinal disorders) | 78 (156) | 26 (35)
Dry mouth (Gastrointestinal disorders) | 9 (10) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 13 (15) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (15) | 2 (2)
Nausea (Gastrointestinal disorders) | 44 (58) | 27 (39)
Stomatitis (Gastrointestinal disorders) | 53 (80) | 27 (37)
Toothache (Gastrointestinal disorders) | 9 (10) | 4 (6)
Vomiting (Gastrointestinal disorders) | 24 (47) | 6 (7)
Asthenia (General disorders) | 25 (39) | 22 (31)
Fatigue (General disorders) | 38 (43) | 21 (22)
Mucosal inflammation (General disorders) | 30 (56) | 16 (21)
Pyrexia (General disorders) | 13 (15) | 13 (16)
COVID-19 (Infections and infestations) | 34 (36) | 16 (17)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 7 (7)
Urinary tract infection (Infections and infestations) | 19 (29) | 12 (14)
Alanine aminotransferase increased (Investigations) | 28 (40) | 21 (29)
Aspartate aminotransferase increased (Investigations) | 28 (35) | 26 (36)
Blood creatinine increased (Investigations) | 9 (16) | 12 (18)
Blood insulin increased (Investigations) | 10 (15) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 13 (16) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (13) | 10 (15)
Neutrophil count decreased (Investigations) | 63 (251) | 64 (210)
Platelet count decreased (Investigations) | 42 (90) | 35 (68)
Weight decreased (Investigations) | 28 (32) | 1 (1)
White blood cell count decreased (Investigations) | 35 (117) | 35 (90)
Decreased appetite (Metabolism and nutrition disorders) | 38 (44) | 14 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 87 (178) | 12 (24)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (14) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (63) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (17) | 20 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 16 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (17) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10) | 9 (12)
Dizziness (Nervous system disorders) | 10 (11) | 13 (15)
Dysgeusia (Nervous system disorders) | 13 (14) | 6 (6)
Headache (Nervous system disorders) | 34 (41) | 22 (28)
Insomnia (Psychiatric disorders) | 16 (17) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 12 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 9 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 30 (30) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (20) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 26 (49) | 21 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04191499/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04191499/SAP_001.pdf